CLINICAL TRIAL: NCT03823911
Title: Cardiovascular Disease in HIV and Hepatitis C: Risk Outcomes After Hepatitis C Eradication
Acronym: CHROME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Poonam Mathur, Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00081300
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases; Hepatitis C; Hiv
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination; ledipasvir, sofosbuvir drug combination; sofosbuvir-velpatasvir drug combination; glecaprevir and pibrentasvir; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- HIV Mono-Infected (Active Comparator): Patients infected with HIV only, and not currently or previously infected with hepatitis C.
  Interventions: Procedure: Cardiac MRI
- Hepatitis C Mono-Infected (Experimental): Patients infected with Hepatitis C and have no evidence of active HIV or hepatitis B infection
  Interventions: Drug: Elbasvir / Grazoprevir Oral Tablet [Zepatier]; Procedure: Cardiac MRI
- HIV and Hepatitis C Co-Infected (Experimental): Patients co-infected with HIV and hepatitis C, and have no evidence of active hepatitis B infection.
  Interventions: Drug: Elbasvir / Grazoprevir Oral Tablet [Zepatier]; Procedure: Cardiac MRI

INTERVENTIONS:
Drug: Elbasvir / Grazoprevir Oral Tablet [Zepatier] — All approved direct-acting antivirals for hepatitis C will be used as the intervention.
  Other Names: Sofosbuvir/Ledipasvir; Sofosbuvir/Velpatasvir; Glecaprevir/Pibrentasvir; Sofosbuvir/Velpatasvir/Voxilaprevir
  Arms: HIV and Hepatitis C Co-Infected; Hepatitis C Mono-Infected
Procedure: Cardiac MRI — Cardiac MRI to assess for myocardial function and fibrosis

SUMMARY:
This is an interventional, non-randomized, controlled prospective study to treat HCV in mono-infected and HIV co-infected individuals and compare cardiovascular risk outcomes to HIV mono-infected controls. This pilot study will demonstrate whether functional cure of HCV reduces myocardial injury and risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or equal to 18 years old
2. Able and willing to sign informed consent
3. Chronically infected with any HCV genotype (1a, 1b, 2, 3, 4, 5, or 6), defined as any individual with documentation of positive HCV antibody and positive HCV RNA test (HCV RNA of 2,000 IU/mL or greater)
4. If HIV+, suppressed on a stable, protocol-approved, ARV regimen for ≥ 8 weeks prior to starting HCV treatment

   1. HIV RNA < 50 copies/mL (or < LLOQ if the local laboratory assay's LLOQ is ≥50 copies/mL) prior to Screening. Subjects with an isolated or unconfirmed HIV RNA > 50 copies/mL (or > LLOQ if the local laboratory assay's LLOQ is ≥50 copies/mL) are not excluded.
   2. CD4 count >100 cells/mm3
5. Willing to have samples stored for future use
6. If tested positive for NS5A resistance-associated polymorphisms or PEG-IFN and ribavirin experienced, able to tolerate ribavirin-containing regimen for 16 weeks. Ribavirin will be administered at the discretion of the PI.
7. Women of childbearing potential who receive ribavirin will have to be willing to commit to abstinence from sexual activity, or use of two forms of contraceptive during treatment and for the 6 months after completion of ribavirin. Men receiving ribavirin who are sexually active with women will also have to be willing to commit to abstinence from sexual activity, or use of two forms of contraceptive during treatment and for the 6 months after completion of ribavirin.

Exclusion Criteria:

1. Decompensated liver disease (Childs Pugh B or C)
2. Unable to comply with research study visits
3. Poor venous access not allowing screening laboratory collection
4. Have any condition that the investigator considers a contraindication to study participation
5. Pregnant or breastfeeding woman
6. Prior HCV treatment with Direct-Acting Antivirals. Note: Patients who are treatment-experienced with PEG-IFN/RBV will not be excluded; their inclusion in the study will be considered by the PI.
7. HIV+ patients with prior HCV treatment who achieved sustained virologic response (SVR)/ functional cure
8. Use of a concomitant medication that is contraindicated with the use of the DAA for HCV treatment (per package insert)
9. Coinfection with HCV and HBV, in partcular HBsAg + patients.

   a. Patients with HBcAb+ will not be excluded, but will have HBV DNA levels checked and will be monitored while on DAA therapy and medically managed as considered appropriate by the PI.
10. Have any condition that the investigator considers a contraindication to study participation or not eligible per standard of care for HCV treatment
11. Patients with the following devices are excluded from participating in the cardiovascular MRI study:

    * Central nervous system aneurysm clip
    * Implanted neural stimulator
    * Implanted cardiac pacemaker or defibrillator
    * Cochlear implant
    * Ocular foreign body (e.g. metal shavings)
    * Implanted insulin pump
    * Metal shrapnel or bullet
12. The following groups of people are also excluded from participating in the cardiovascular MRI study:

    * Patients with stable renal disease (estimated glomerular filtration rate (eGFR)<30ml/min/1.73m2 body surface area. The eGFR must be within two weeks of the the MRI exam.
    * Patients with acute renal disease.
13. Patients who choose to have the cardiac MRI and are over 60 years of age, have a history of renal failure, or have type I or II diabetes mellitus must have laboratory tests the same day as the MRI exam.
14. Positive urine drug screen at screening. Not all patients with positive drug screen will be excluded; decision will be made by the PI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poonam Mathur, DO, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Unity Parkside Health Center, Washington D.C., District of Columbia
  - Institute of Human Virology, CRU, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Stored samples will be sent to the Institute of Human Virology at the University of Maryland and to BHF Centre for Cardiovascular Sciences:
  Individuals with new seroconversion to HIV will have samples sent for viral sequencing and phylogenetic analysis. Individuals with detectable HCV RNA after completion of HCV treatment or new infection during the follow up period will have current sample, and baseline stored sample sent for viral sequencing and phylogenetic analysis.
  In addition, we will study the viral and host immunity to HCV and HIV in all patients. The results will be used to characterize each individual with regards to immune status and chronicity of disease.
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV Mono-Infected | Hepatitis C Mono-Infected | HIV and Hepatitis C Co-Infected
Started | 43 | 37 | 7
Completed | 29 | 24 | 1
Not Completed | 14 | 13 | 6
Not completed — Lost to Follow-up | 1 | 5 | 2
Not completed — Did not meet eligibility criteria | 13 | 7 | 4
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Mono-Infected | Hepatitis C Mono-Infected | HIV and Hepatitis C Co-Infected | Total
Number analyzed (Participants) | 43 | 37 | 7 | 87
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 78] | 58 [26 to 71] | 56 [34 to 67] | 55 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 1 | 37
  Male | 24 | 20 | 6 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 37 | 32 | 6 | 75
  White | 4 | 3 | 1 | 8
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 37 | 7 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiovascular Disease Risk From Baseline to After Functional Cure of Hepatitis C, as Measured by High-sensitivity C-reactive Protein
Description: Change in high-sensitivity C-reactive protein
Time Frame: Baseline to 72 weeks after functional cure of HCV
Population: 13 participants were analyzed in the hepatitis C mono-infected group and 1 participant in the HIV-HCV co-infected group since other participants were lost to follow-up and week 72 data was available for these participants only.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Hepatitis C Mono-Infected | HIV and Hepatitis C Co-Infected
Number analyzed (Participants) | 13 | 1
mg/L | 0.6 (0.96) | 0 (0)

2. Secondary Outcome: Change in Troponin I and Troponin T From Baseline to After Functional Cure of Hepatitis C
Description: Change in the cardiac biomarkers Troponin I and Troponin T
Time Frame: Baseline to 48 weeks after functional cure of HCV
Population: Data on troponin I and T were not collected for any of the participants, therefore the outcome cannot be reported
Arm/Group | Hepatitis C Mono-Infected | HIV and Hepatitis C Co-Infected
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 12 weeks while on hepatitis C therapy
Arm/Group | HIV Mono-Infected | Hepatitis C Mono-Infected | HIV and Hepatitis C Co-Infected
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/37 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/37 | 0/7
Other Adverse Events (participants affected / at risk) | 0/43 | 0/37 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03823911/Prot_SAP_000.pdf